CLINICAL TRIAL: NCT01068366
Title: Nickel Allergy With Septal Occluder Using Amplatzer and Helex Devices (NASAH) Trial
Brief Title: Nickel Allergy With Septal Closure Devices
Acronym: NASAH
Status: Terminated | Type: Observational
Why Stopped: PI re-located.
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 38813
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Atrial Septal Defect; Patent Foramen Ovale; Allergic Reaction to Nickel
Keywords: Nickel Allergic Syndrome; Septal Closure Devices
MeSH Terms: conditions — Heart Septal Defects, Atrial; Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is for patients who have been diagnosed with either a Patent Foramen Ovale [PFO] or an Atrial Septal Defect [ASD]. These are a type of hole located in the wall that separates the top two (2) chambers of the heart. You have been recommended to receive an atrial septal occluder device [a device specifically designed to close PFOs and ASDs] implanted in your heart to close this hole. Because these devices are made of materials that contain nickel, this trial is being conducted to perform blood nickel tests on those patients already referred for an atrial septal occluder device such as yourself. The purpose of this study is to compare levels of nickel in the blood in patients receiving either the Amplatzer or the Helex devices.

DETAILED DESCRIPTION:
This is a single-center, single-operator, investigator-initiated, investigator-funded, open-label, non-randomized cohort study. Inclusion criteria include patients ≥18 years, secundum atrial septal defect (ASD) ≤1cm on transesophageal echocardiography or patent foramen ovale (PFO), without contraindications to antiplatelet and/or antithrombotic therapy, and suitable anatomy for device closure with one of the following: Amplatzer atrial septal occluder, Amplatzer Cribriform septal occluder, Amplatzer PFO occluder, or the Gore Helex septal occluder. After device implantation, routine clinical followup will be performed, including transthoracic echocardiography at 1 day, 1 month, and 6 months, and 48-Holter monitoring for arrhythmia at 1 month.

Research related study procedures are blood draws to measure nickel levels and a patient questionnaire about symptoms. Blood draws will be done at baseline [from the femoral venous sheath immediately prior to device implantation] and at one (1) day, one (1) month, three (3) months and six (6) months. The Questionnaire will be completed at one (1) month, three (3) months and six (6) months but can be done over the telephone if patient is having blood drawn at a lab closer to their home. Patient participation is complete after collection of the 6 month blood results and patient questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years,
* Secundum atrial septal defect (ASD) ≤ 1 cm on transesophageal echocardiography or patent foramen ovale (PFO), without contraindications to antiplatelet and/or antithrombotic therapy, and
* Suitable anatomy for device closure with one of the following: Amplatzer atrial septal occluder, Amplatzer Cribriform septal occluder, Amplatzer PFO occluder, or the Gore Helex septal occluder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already scheduled for ASD or PFO closure with Amplatzer or Helex devices.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The difference in serum nickel levels | 1 month post device implantation

SECONDARY OUTCOMES:
Device allergic syndrome | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D. Michaels, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States